CLINICAL TRIAL: NCT03055195
Title: Study 205050: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Mepolizumab Administered Subcutaneously in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of Mepolizumab in Subjects With Moderate to Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study reached pre-determined futility criteria following interim analysis. No safety concerns were noted.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205050
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2017-02-13; First posted 2017-02-16 (Actual); Results first posted 2018-12-26 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Dermatitis, Atopic
Keywords: subcutaneous; safety; mepolizumab; efficacy; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab (Experimental): Eligible subjects will receive mepolizumab 100 mg subcutaneously every 4 weeks on Day 1, Week 4, Week 8, and Week 12
  Interventions: Drug: Mepolizumab 100 mg
- Placebo (Placebo Comparator): Eligible subjects will receive matching placebo subcutaneously every 4 weeks on Day 1, Week 4, Week 8, and Week 12
  Interventions: Drug: Placebo matching mepolizumab

INTERVENTIONS:
Drug: Mepolizumab 100 mg — Mepolizumab is available as lyophilized powder in sterile vials for injection. The content is reconstituted with 1.2 milliliter (mL) Sterile Water just prior to use. Subjects will receive 1mL (100 mg/mL) bolus subcutaneous injections.
  Arms: Mepolizumab
Drug: Placebo matching mepolizumab — Placebo is available as 0.9% sodium chloride solution. Subjects will receive 1mL bolus subcutaneous injections.
  Arms: Placebo

SUMMARY:
Mepolizumab is a humanized Immunoglobulin G1 (IgG1) monoclonal antibody (mAb) that acts on Interleukin-5 (IL-5), which is responsible for the growth and differentiation, recruitment, activation, and survival of eosinophils; thereby reducing the production and survival of eosinophils which may be therapeutic in subjects with atopic dermatitis (AD). This study will investigate the efficacy and safety of mepolizumab (100 milligram [mg] subcutaneous [SC] administered every 4 weeks) compared with placebo in adult subjects with moderate to severe atopic dermatitis (AD). Subjects will be randomized 1:1 to either placebo SC or mepolizumab SC. The study will comprise of a pre-screening period of up to approximately 4 weeks, a screening period of up to 2 weeks, followed by a 16-Week study treatment period (16 weeks with the last dose of study treatment at Week 12) and follow-up period of up to 4-week. The total duration of subject participation will be approximately 26 weeks. (Note: For subjects, who may need to stop treatment with a biologic, the total Pre-Screening and Screening period may last up to 20 weeks and total duration of participation in the study may be up to 40 weeks).

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* AD diagnosed by the Eichenfield revised criteria of Hanifin and Rajka.
* Diagnosis of AD >=2 years prior to the Screening visit.
* An IGA score >=3 at the Screening and Baseline visits.
* AD involvement of >=10% body surface area at the Screening and Baseline visits.
* EASI score >=16 at the Screening and Baseline visits.
* Absolute blood eosinophil count >=350 cells/microliter at the Screening visit.
* Applied the same non-prescription, non-medicated (without an active ingredient) emollient twice daily for at least 7 days immediately before the Baseline visit.
* Recent history (<=6 months prior to the Screening visit) of inadequate response to a stable regimen of prescription topical medication or for whom prescription topical medications are not tolerated or where there is a concern for potential side effects, such as skin thinning or increased risk of hypothalamic-pituitary-adrenal [HPA] suppression; as well as, inadequate response to optimization of non-pharmacological measures such as moisturizers. Inadequate response to a stable regimen of prescription topical medication (such as medium to high potency topical corticosteroids or topical calcineurin inhibitors) is defined as failure to achieve and maintain remission or low disease activity state (equivalent to an IGA score =0 [clear] to 2 [mild]) despite treatment for the recommended duration as per label or for the maximum duration recommended for the subject treatment, whichever is shorter.
* Male or female: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions: Non-reproductive potential- Pre-menopausal females with documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy; and postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 16 weeks after the last dose of study medication.
* The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Subject is able to give signed informed consent that includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria

* Other types of eczema.
* Any other concomitant skin disorder (e.g., generalized erythroderma such as Netherton's Syndrome, or psoriasis), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of AD lesions or compromise subject safety.
* Immunocompromised (e.g., lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich Syndrome) or has a history of malignant disease within 5 years before the Baseline visit. Note: Subjects with successfully treated basal cell carcinoma (no more than 3 lesions), squamous cell carcinoma of the skin, or cervical carcinoma in situ, with no evidence of recurrence within the 3 years prior to the Baseline visit may participate in the study.
* A positive history for human immunodeficiency virus (HIV) antibody.
* Chronic or acute infection requiring treatment with oral or intravenous (IV) antibiotics, antivirals, anti-protozoals, or antifungals within 4 weeks before the Screening visit or anytime between the Screening and Baseline visits.
* Superficial skin infections within 1 week before the Screening visit.
* Known, pre-existing or suspected parasitic infection within 6 months before the Screening visit.
* Other known or suspected conditions that could lead to elevated eosinophils, for example, hypereosinophilic syndromes including eosinophilic granulomatosis with polyangiitis (EGPA, also known as Churg-Strauss Syndrome), eosinophilic esophagitis, or severe asthma.
* A history or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, may interfere with the subject's completion of the study.
* ALT >2x upper limit of normal (ULN)
* Bilirubin >1.5x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT Interval Corrected by Fridericia Correction Formula (QTcF) >450 milliseconds (msec) or QTcF >480 msec in subjects with Bundle Branch Block.
* Clinically significant abnormality in the hematological or biochemical screen, as judged by the investigator.
* Previously treated with mepolizumab or participated in a previous mepolizumab clinical study.
* Prior treatment with any of the medications or treatments listed in Table 1 within the indicated periods before the Screening visit.
* Prolonged exposure to natural (e.g, sunlight) ultraviolet (UV) radiation within 4 weeks prior to the Baseline visit and/or intention to have such exposure during the study, which is thought by the investigator to potentially impact the subject's AD.
* More than 2 visits per week to a tanning booth or parlor in the 4 weeks prior to the Baseline visit.
* Onset of a new exercise routine or major change to a previous exercise routine within 2 weeks before randomization, or unwilling to maintain current level of physical activity throughout the length of participation in this study.
* History of alcohol or other substance abuse within the last 2 years.
* Hypersensitivity to mepolizumab or any of its excipients.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the Baseline visit.
* Subject is a member of the investigational team or his/her immediate family.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (11):
  - GSK Investigational Site, Fort Smith, Arkansas
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Sandy Springs, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Norfolk, Virginia
- Canada (9):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20100

REFERENCES:
- [Background] Kang EG, Narayana PK, Pouliquen IJ, Lopez MC, Ferreira-Cornwell MC, Getsy JA. Efficacy and safety of mepolizumab administered subcutaneously for moderate to severe atopic dermatitis. Allergy. 2020 Apr;75(4):950-953. doi: 10.1111/all.14050. Epub 2019 Oct 9. No abstract available. PMID 31515809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study investigated the efficacy and safety of mepolizumab administered subcutaneously (SC) in adults with moderate to severe atopic dermatitis. A total of 34 participants were enrolled at different centers in Canada and United States.
Pre-assignment Details: This study was terminated early, as this study reached pre-determined futility criteria following interim analysis.
Groups:
- Placebo SC: Participants received placebo (0.9 percent sodium chloride solution) SC injection administered into the upper arm, abdomen, or thigh every 4 weeks.
- Mepolizumab 100 mg SC: Participants received 100 milligram (mg) of Mepolizumab SC injection administered into the upper arm, abdomen, or thigh every 4 weeks.
Period: Overall Study
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Started | 16 | 18
Completed | 4 | 4
Not Completed | 12 | 14
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Study Terminated by Sponsor | 2 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC | Mepolizumab 100 mg SC | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.8 (9.95) | 34.6 (13.99) | 32.8 (12.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 9 | 12 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 1 | 1 | 2
  Asian - East Asian Heritage | 5 | 4 | 9
  Asian - Japanese Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 2 | 2 | 4
  Black Or African American | 2 | 1 | 3
  White - White/Caucasian/European Heritage | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator's Global Assessment (IGA) Score of 0 or 1 and at Least a 2- Grade Improvement at Week 16
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's atopic dermatitis . It is a static 5-point morphological assessment of overall disease severity determined by the investigator, sub-investigator, or trained healthcare professional with required qualifications on a scale of 0 to 4 where, 0-clear, 1-almost clear, 2-mild, 3-moderate, and 4- severe. Higher score indicates severity of disease. A responder is defined as a participant who had an IGA score of 0 or 1 and a minimum 2-grade improvement from Baseline. Number of participants with IGA score of 0 or 1 and at least a 2- grade improvement at Week 16 was presented.
Time Frame: Week 16
Population: Intent-to-Treat Population comprised of all participants who were randomized and who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 16 | 18
Participants | 0 | 2
Statistical Analysis 1: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportions Difference = 11, 90% CI 2-sided [-1.1 to 23.3] — Difference in Proportions between Mepolizumab 100 mg SC versus Placebo SC has been presented

2. Secondary Outcome: Mean Percentage Change in Eczema Area and Severity Index (EASI) Score From Baseline to Each Study Visit
Description: EASI scoring system is a standardized clinical tool for the assessment of atopic dermatitis that takes into account overall extent of the percent body surface area (% BSA) involved and severity scores for each clinical signs (erythema, induration/papulation, excoriation, and lichenification). Severity scores were graded on a 4-point scale, 0(absent) to 3(severe) for each body regions (head and neck, upper extremities, lower extremities, and trunk). The severity scores for each signs were summed for each region and multiplied by the % BSA area score and by the appropriate proportionality multiplier (for participants >=8 years of age, 0.1 for head, 0.2 upper extremities, 0.3 for trunk and 0.4 for lower extremities) to generate a regional EASI score. The regional EASI scores were then summed to yield the final EASI score. Baseline is defined as latest pre-dose assessment. Percent change from Baseline is Post-Baseline Visit Value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: Intent-to-Treat Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 16 | 18
Percent change
  Week 4, n=16, 17: number analyzed (Participants) | 16 | 17
  Week 4, n=16, 17 | -22.508 (30.2511) | -24.556 (45.4823)
  Week 8,n=15, 16: number analyzed (Participants) | 15 | 16
  Week 8,n=15, 16 | -30.497 (29.0671) | -43.904 (43.4749)
  Week 12, n= 11, 11: number analyzed (Participants) | 11 | 11
  Week 12, n= 11, 11 | -22.372 (31.7156) | -42.464 (49.2445)
  Week 16, n=8, 6: number analyzed (Participants) | 8 | 6
  Week 16, n=8, 6 | -32.269 (27.8121) | -31.921 (50.0658)
  Week 20, n=4, 4: number analyzed (Participants) | 4 | 4
  Week 20, n=4, 4 | 1.327 (32.5577) | -63.938 (34.2710)

3. Secondary Outcome: Number of Participants With an IGA Score of 0 or 1 and at Least a 2-grade Improvement at Each Study Visit
Description: The IGA is a clinical tool for assessing the current state/severity of a participant's atopic dermatitis . It is a static 5-point morphological assessment of overall disease severity determined by the investigator, sub-investigator, or trained healthcare professional with required qualifications on a scale of 0 to 4 where, 0-clear, 1-almost clear, 2-mild, 3-moderate, and 4- severe. Higher score indicates severity of disease. A Responder is defined as a participant who had an IGA score of 0 or 1 and a minimum 2-grade improvement from Baseline. Participants withdrawn early from the study were assigned to be a non-responder for all weeks after withdrawal. Number of participants with IGA score of 0 or 1 and at least a 2- grade improvement at each study visit (Weeks 4, 8, 12, 16 and 20) is presented.
Time Frame: Weeks 4, 8, 12, 16 and 20
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 16 | 18
Participants
  Week 4 | 1 | 1
  Week 8 | 0 | 2
  Week 12 | 0 | 2
  Week 16 | 0 | 2
  Week 20 | 0 | 1
Statistical Analysis 1: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportion Difference = -1, 90% CI 2-sided [-14.0 to 12.6] — Difference in Proportions between Mepolizumab 100 mg SC Versus Placebo SC at Week 4 has been presented
Statistical Analysis 2: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportion Difference = 11, 90% CI 2-sided [-1.1 to 23.3] — Difference in Proportions between Mepolizumab 100 mg SC Versus Placebo SC at Week 8 has been presented
Statistical Analysis 3: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportion Difference = 11, 90% CI 2-sided [-1.1 to 23.3] — Difference in Proportions between Mepolizumab 100 mg SC Versus Placebo SC at Week 12 has been presented
Statistical Analysis 4: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportion Difference = 11, 90% CI 2-sided [-1.1 to 23.3] — Difference in Proportions between Mepolizumab 100 mg SC Versus Placebo SC at Week 16 has been presented
Statistical Analysis 5: Comparison: Placebo SC vs Mepolizumab 100 mg SC; Test type: Other; Proportion Difference = 6, 90% CI 2-sided [-3.3 to 14.4] — Difference in Proportions between Mepolizumab 100 mg SC Versus Placebo SC at Week 20 has been presented

4. Secondary Outcome: Number of Participants With On-treatment Adverse Events (AEs), Serious Adverse Events (SAEs) and Non-serious Adverse Events (nSAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. On-treatment AES were reported on or after treatment start date and on or before treatment stop date (plus 28 days). Number of participants with AEs, SAEs and nSAEs is presented.
Time Frame: Up to Week 20
Population: Safety Population comprised of all participants who received at least one dose of a study treatment. One participant from Placebo arm received Mepolizumab at Day 1 instead of placebo due to error.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Participants
  Any AE | 7 | 1
  Any SAE | 0 | 0
  Any nSAE | 7 | 1

5. Secondary Outcome: Number of Participants With On-treatment AEs of Special Interest Reported as Local Site Injection Reaction and Systemic Reactions
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with local site injection reaction and systemic reactions were reported.
Time Frame: Up to Week 20
Population: Safety Population. One participant from Placebo arm received Mepolizumab at Day 1 instead of placebo due to error.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Participants
  Local site injection reaction | 0 | 0
  Systemic reaction | 0 | 0

6. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). One participant from Placebo arm received Mepolizumab at Day 1 instead of placebo due to error.
Measure: Mean (Standard Deviation); unit: Billion cells per liter (10^9/L)
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Billion cells per liter (10^9/L)
  Basophils, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Basophils, Week 4, n=15,17 | 0.000 (0.0146) | -0.021 (0.0293)
  Basophils, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Basophils, Week 8, n=12,17 | 0.013 (0.0234) | -0.018 (0.0282)
  Basophils, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Basophils, Week 12, n=10,11 | 0.007 (0.0164) | -0.010 (0.0219)
  Basophils, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Basophils, Week 16, n=7,7 | -0.006 (0.0190) | -0.001 (0.0195)
  Basophils, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Basophils, Week 20, n=3,4 | 0.000 (0.0100) | -0.008 (0.0150)
  Eosinophils, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Eosinophils, Week 4, n=15,17 | -0.028 (0.5179) | -0.567 (0.2498)
  Eosinophils, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Eosinophils, Week 8, n=12,17 | -0.193 (0.3991) | -0.601 (0.2820)
  Eosinophils, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Eosinophils, Week 12, n=10,11 | -0.086 (0.2866) | -0.605 (0.3668)
  Eosinophils, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Eosinophils, Week 16, n=7,7 | 0.000 (0.3354) | -0.517 (0.4007)
  Eosinophils, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Eosinophils, Week 20, n=3,4 | 0.173 (0.7247) | -0.438 (0.3721)
  Leukocytes, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Leukocytes, Week 4, n=15,17 | -0.01 (1.307) | -0.75 (1.471)
  Leukocytes, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Leukocytes, Week 8, n=12,17 | -0.23 (1.393) | -0.77 (1.162)
  Leukocytes, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Leukocytes, Week 12, n=10,11 | 0.68 (1.466) | -0.59 (2.257)
  Leukocytes, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Leukocytes, Week 16, n=7,7 | 0.37 (1.053) | -0.44 (1.427)
  Leukocytes, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Leukocytes, Week 20, n=3,4 | -0.10 (0.866) | -1.12 (1.372)
  Lymphocytes, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Lymphocytes, Week 4, n=15,17 | 0.001 (0.3654) | -0.104 (0.4309)
  Lymphocytes, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Lymphocytes, Week 8, n=12,17 | 0.046 (0.5113) | -0.140 (0.4461)
  Lymphocytes, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Lymphocytes, Week 12, n=10,11 | -0.127 (0.5121) | -0.057 (0.3453)
  Lymphocytes, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Lymphocytes, Week 16, n=7,7 | 0.409 (0.8914) | -0.051 (0.2543)
  Lymphocytes, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Lymphocytes, Week 20, n=3,4 | 0.240 (0.4251) | -0.095 (0.1638)
  Monocytes, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Monocytes, Week 4, n=15,17 | 0.057 (0.1247) | -0.011 (0.1508)
  Monocytes, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Monocytes, Week 8, n=12,17 | 0.028 (0.1207) | -0.090 (0.1634)
  Monocytes, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Monocytes, Week 12, n=10,11 | 0.029 (0.1347) | -0.070 (0.1532)
  Monocytes, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Monocytes, Week 16, n=7,7 | 0.039 (0.1206) | 0.017 (0.0939)
  Monocytes, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Monocytes, Week 20, n=3,4 | 0.073 (0.2641) | 0.010 (0.1268)
  Neutrophils, Week 4, n=15,17: number analyzed (Participants) | 15 | 17
  Neutrophils, Week 4, n=15,17 | -0.029 (1.2133) | -0.062 (1.3958)
  Neutrophils, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Neutrophils, Week 8, n=12,17 | -0.103 (1.3031) | 0.068 (0.8773)
  Neutrophils, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Neutrophils, Week 12, n=10,11 | 0.864 (1.8011) | 0.130 (1.9898)
  Neutrophils, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Neutrophils, Week 16, n=7,7 | -0.089 (1.2211) | 0.104 (1.0966)
  Neutrophils, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Neutrophils, Week 20, n=3,4 | -0.577 (0.5387) | -0.587 (1.3189)
  Platelets, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Platelets, Week 4, n=15,18 | 2.6 (30.86) | -4.8 (35.02)
  Platelets, Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Platelets, Week 8, n=12,17 | 1.3 (45.31) | 7.5 (36.83)
  Platelets, Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Platelets, Week 12, n=10,11 | -4.5 (36.92) | -16.8 (23.34)
  Platelets, Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Platelets, Week 16, n=7,7 | 1.4 (29.73) | -27.7 (38.87)
  Platelets, Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Platelets, Week 20, n=3,4 | 11.3 (15.57) | -14.0 (35.07)

7. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Picograms
  Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  Week 4,n=15,18 | 0.05 (0.582) | 0.13 (0.407)
  Week 8,n=12,17: number analyzed (Participants) | 12 | 17
  Week 8,n=12,17 | -0.08 (0.564) | 0.09 (0.578)
  Week 12,n=10,11: number analyzed (Participants) | 10 | 11
  Week 12,n=10,11 | 0.08 (0.461) | 0.15 (0.670)
  Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  Week 16,n=7,7 | 0.46 (0.336) | 0.11 (0.708)
  Week 20,n=3,4: number analyzed (Participants) | 3 | 4
  Week 20,n=3,4 | 0.33 (0.252) | 0.55 (0.926)

8. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Femtoliter
  Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  Week 4,n=15,18 | 0.2 (2.08) | 0.3 (2.45)
  Week 8,n=12,17: number analyzed (Participants) | 12 | 17
  Week 8,n=12,17 | -0.4 (1.56) | -0.4 (2.58)
  Week 12,n=10,11: number analyzed (Participants) | 10 | 11
  Week 12,n=10,11 | -1.1 (1.60) | -0.7 (2.90)
  Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  Week 16,n=7,7 | -0.7 (0.76) | -1.7 (3.25)
  Week 20,n=3,4: number analyzed (Participants) | 3 | 4
  Week 20,n=3,4 | -0.3 (1.53) | 0.3 (2.63)

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Trillion cells/liter (10^12 cell/L)
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Trillion cells/liter (10^12 cell/L)
  Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Week 4, n=15,18 | 0.02 (0.262) | 0.01 (0.226)
  Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Week 8, n=12,17 | 0.06 (0.294) | -0.02 (0.283)
  Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Week 12, n=10,11 | 0.08 (0.210) | 0.06 (0.234)
  Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Week 16, n=7,7 | -0.01 (0.204) | 0.10 (0.153)
  Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Week 20, n=3,4 | 0.13 (0.252) | 0.07 (0.096)

10. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: Hematocrit. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Percentage of red blood cells in blood
  Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Week 4, n=15,18 | 0.0030 (0.02071) | 0.0021 (0.02555)
  Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Week 8, n=12,17 | 0.0024 (0.02171) | -0.0042 (0.02357)
  Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Week 12, n=10,11 | 0.0011 (0.01813) | 0.0005 (0.01873)
  Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Week 16, n=7,7 | -0.0057 (0.01616) | 0.0007 (0.01701)
  Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Week 20, n=3,4 | 0.0130 (0.01400) | 0.0082 (0.00967)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Hemoglobin. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Grams per liter
  Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Week 4, n=15,18 | 1.0 (7.29) | 0.9 (6.82)
  Week 8, n=12,17: number analyzed (Participants) | 12 | 17
  Week 8, n=12,17 | 1.0 (7.48) | 0.0 (6.76)
  Week 12, n=10,11: number analyzed (Participants) | 10 | 11
  Week 12, n=10,11 | 2.6 (5.44) | 2.3 (5.55)
  Week 16, n=7,7: number analyzed (Participants) | 7 | 7
  Week 16, n=7,7 | 1.7 (6.32) | 3.7 (4.19)
  Week 20, n=3,4: number analyzed (Participants) | 3 | 4
  Week 20, n=3,4 | 6.7 (6.51) | 5.0 (2.45)

12. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP and AST . Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
International units per liter (IU/L)
  ALT, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  ALT, Week 4, n=15,18 | 1.4 (5.45) | 0.3 (27.10)
  ALT, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  ALT, Week 8, n=11,16 | 5.9 (22.31) | -6.3 (21.96)
  ALT, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  ALT, Week 12, n=7,11 | -2.0 (10.00) | -3.5 (11.01)
  ALT, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  ALT, Week 16, n=5,7 | 2.4 (6.69) | 1.7 (8.40)
  ALP, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  ALP, Week 4, n=15,18 | -2.3 (5.85) | -1.9 (10.06)
  ALP, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  ALP, Week 8, n=11,16 | 0.3 (6.89) | 0.4 (13.86)
  ALP, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  ALP, Week 12, n=7,11 | 3.9 (3.85) | -3.8 (7.43)
  ALP, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  ALP, Week 16, n=5,7 | 3.2 (7.26) | -2.6 (6.48)
  AST, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  AST, Week 4, n=15,18 | 0.6 (4.00) | -3.0 (11.60)
  AST, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  AST, Week 8, n=11,16 | -0.1 (8.87) | -4.9 (11.11)
  AST, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  AST, Week 12, n=7,11 | -2.1 (5.27) | -6.0 (13.34)
  AST, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  AST, Week 16, n=5,7 | 0.4 (5.13) | -1.0 (8.64)

13. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected to analyze the chemistry parameters: Albumin and Protein. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Grams per liter
  Albumin, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Albumin, Week 4, n=15,18 | -0.5 (2.75) | 0.3 (3.31)
  Albumin, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Albumin, Week 8, n=11,16 | -0.6 (2.42) | 0.7 (3.46)
  Albumin, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Albumin, Week 12, n=7,11 | -0.6 (2.23) | 1.1 (2.77)
  Albumin, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Albumin, Week 16, n=5,7 | -1.4 (3.13) | 1.9 (1.86)
  Protein, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Protein, Week 4, n=15,18 | -0.5 (3.02) | 1.3 (3.41)
  Protein, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Protein, Week 8, n=11,16 | 0.8 (4.02) | 1.6 (4.59)
  Protein, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Protein, Week 12, n=7,11 | 0.4 (2.70) | 1.6 (2.54)
  Protein, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Protein, Week 16, n=5,7 | -1.2 (4.32) | 2.7 (3.64)

14. Secondary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine, Direct Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: Bilirubin, Creatinine and Direct Bilirubin. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Micromoles per liter
  Bilirubin, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Bilirubin, Week 4, n=15,18 | 1.2 (3.53) | 2.0 (3.82)
  Bilirubin, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Bilirubin, Week 8, n=11,16 | -0.4 (3.32) | 1.6 (4.27)
  Bilirubin, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Bilirubin, Week 12, n=7,11 | -0.9 (2.54) | 0.7 (3.93)
  Bilirubin, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Bilirubin, Week 16, n=5,7 | -1.2 (1.79) | 2.3 (5.59)
  Creatinine, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Creatinine, Week 4, n=15,18 | 2.77 (10.027) | 0.74 (8.097)
  Creatinine, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Creatinine, Week 8, n=11,16 | 0.74 (7.250) | -0.81 (5.150)
  Creatinine, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Creatinine, Week 12, n=7,11 | 0.63 (2.799) | 1.62 (6.693)
  Creatinine, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Creatinine, Week 16, n=5,7 | 1.24 (5.379) | -1.63 (11.755)
  Direct Bilirubin, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Direct Bilirubin, Week 4, n=15,18 | 0.3 (1.28) | 0.2 (1.17)
  Direct Bilirubin, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Direct Bilirubin, Week 8, n=11,16 | -0.5 (1.29) | 0.0 (1.26)
  Direct Bilirubin, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Direct Bilirubin, Week 12, n=7,11 | -0.6 (0.98) | 0.2 (1.08)
  Direct Bilirubin, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Direct Bilirubin, Week 16, n=5,7 | 0.0 (0.00) | 0.3 (0.76)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium and Urea
Description: Blood samples were collected to analyze the chemistry parameters: Calcium, Glucose, Potassium, Sodium and Urea. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, and 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Millimoles per liter (mmol/L)
  Calcium, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Calcium, Week 4, n=15,18 | -0.003 (0.0692) | -0.004 (0.1130)
  Calcium, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Calcium, Week 8, n=11,16 | 0.007 (0.1093) | 0.001 (0.1097)
  Calcium, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Calcium, Week 12, n=7,11 | 0.031 (0.1232) | -0.005 (0.1110)
  Calcium, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Calcium, Week 16, n=5,7 | -0.076 (0.1126) | 0.043 (0.0941)
  Glucose, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Glucose, Week 4, n=15,18 | -0.13 (0.841) | 0.20 (0.707)
  Glucose, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Glucose, Week 8, n=11,16 | -0.56 (1.267) | 0.53 (0.846)
  Glucose, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Glucose, Week 12, n=7,11 | 0.90 (2.653) | 0.14 (1.002)
  Glucose, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Glucose, Week 16, n=5,7 | 0.26 (0.783) | 0.21 (0.857)
  Potassium, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Potassium, Week 4, n=15,18 | -0.02 (0.265) | -0.01 (0.252)
  Potassium, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Potassium, Week 8, n=11,16 | 0.07 (0.290) | -0.03 (0.272)
  Potassium, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Potassium, Week 12, n=7,11 | 0.19 (0.254) | -0.06 (0.191)
  Potassium, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Potassium, Week 16, n=5,7 | 0.04 (0.288) | -0.09 (0.363)
  Sodium, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Sodium, Week 4, n=15,18 | 0.3 (1.88) | -0.9 (1.94)
  Sodium, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Sodium, Week 8, n=11,16 | 1.0 (1.34) | -0.2 (1.76)
  Sodium, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Sodium, Week 12, n=7,11 | 0.0 (1.83) | 0.1 (1.04)
  Sodium, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Sodium, Week 16, n=5,7 | -1.2 (1.30) | 0.4 (2.30)
  Urea, Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  Urea, Week 4, n=15,18 | 0.23 (1.015) | -0.25 (1.204)
  Urea, Week 8, n=11,16: number analyzed (Participants) | 11 | 16
  Urea, Week 8, n=11,16 | 0.41 (1.114) | -0.78 (1.722)
  Urea, Week 12, n=7,11: number analyzed (Participants) | 7 | 11
  Urea, Week 12, n=7,11 | -0.07 (1.813) | -0.59 (1.998)
  Urea, Week 16, n=5,7: number analyzed (Participants) | 5 | 7
  Urea, Week 16, n=5,7 | 0.30 (1.304) | -0.50 (2.255)

16. Secondary Outcome: Number of Participants With Worst Post Baseline Potential Clinical Importance (PCI) Value for Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; hematocrit, hemoglobin, leukocytes and platelets. PCI ranges were < 0.201 or >0.599 proportion of red blood cells in blood for hematocrit, <71 or >199 grams per liter for hemoglobin, <31 or >1499 Giga cells per liter for platelets and for leukocytes < 1.1 Giga cells per liter. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants with laboratory value category "To Low" and "To High" were presented. Only those parameters having worst post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to Week 20
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. One participant from Placebo arm received Mepolizumab at Day 1 instead of placebo due to error.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 18
Participants
  Hematocrit, To Low | 0 | 0
  Hematocrit, To High | 0 | 0
  Hemoglobin, To Low | 0 | 0
  Hemoglobin, To High | 0 | 0
  Leukocytes, To Low | 0 | 0
  Leukocytes, To High | 0 | 0
  Platelets, To Low | 0 | 0
  Platelets, To High | 0 | 0

17. Secondary Outcome: Number of Participants With Worst Post Baseline PCI Value for Chemistry Parameters
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: ALT, Calcium, glucose, Potassium and sodium. PCI ranges were >143 units per liter (U/L) for ALT (Age category: 3-12 years) and >239 U/L for ALT (Age category: 13+ years), <1.50 or >3.24 mmol/L for calcium, < 2.2 or > 27.8 mmol/L for glucose, <2.8 or >6.5 mmoL/L for potassium , and <120 or >160 mmoL/L for sodium. Participants were counted in the worst case category that their value changes to (low, normal , or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Only those parameters having worst post-Baseline PCI values were presented. Day 1 was considered as Baseline.
Time Frame: Up to Week 16
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 18
Participants
  ALT, To Low | 0 | 0
  ALT, To High | 0 | 0
  Calcium, To Low | 0 | 0
  Calcium, To High | 0 | 0
  Glucose, To Low | 0 | 0
  Glucose, To High | 0 | 0
  Potassium, To Low | 0 | 0
  Potassium, To High | 0 | 0
  Sodium, To Low | 0 | 0
  Sodium, To High | 0 | 0

18. Secondary Outcome: Change From Baseline in PR Interval, QRS Duration, QT Interval and QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF)
Description: Triplicate 12-lead electrocardiograms (ECG) were obtained to measure PR Interval, QRS Duration, QT Interval and QTcF Interval. Screening was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Screening) and Weeks 4, 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Milliseconds
  PR Interval; Week 4, n=15,18: number analyzed (Participants) | 15 | 18
  PR Interval; Week 4, n=15,18 | 9.1 (9.91) | -0.5 (10.62)
  PR Interval; Week 16,n=12,16: number analyzed (Participants) | 12 | 16
  PR Interval; Week 16,n=12,16 | -1.3 (15.43) | 1.5 (12.54)
  QRS duration; Week 4; n=15,18: number analyzed (Participants) | 15 | 18
  QRS duration; Week 4; n=15,18 | -0.9 (5.93) | 3.1 (7.71)
  QRS duration; Week 16,n=12,16: number analyzed (Participants) | 12 | 16
  QRS duration; Week 16,n=12,16 | -2.2 (6.51) | 0.9 (8.27)
  QT Interval; Week 4; n=15,18: number analyzed (Participants) | 15 | 18
  QT Interval; Week 4; n=15,18 | -5.8 (17.65) | -4.7 (16.32)
  QT Interval; Week 16,n=12,16: number analyzed (Participants) | 12 | 16
  QT Interval; Week 16,n=12,16 | -10.8 (18.05) | -4.1 (23.42)
  QTc F Interval; Week 4; n=15,18: number analyzed (Participants) | 15 | 18
  QTc F Interval; Week 4; n=15,18 | -2.4 (11.69) | -6.4 (14.30)
  QTcF Interval; Week 16,n=12,16: number analyzed (Participants) | 12 | 16
  QTcF Interval; Week 16,n=12,16 | -2.1 (18.20) | -5.8 (17.68)

19. Secondary Outcome: Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Millimeters of mercury (mmHg)
  DBP, Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  DBP, Week 4,n=15,18 | 1.3 (8.22) | 4.5 (9.73)
  DBP, Week 8,n=14,17: number analyzed (Participants) | 14 | 17
  DBP, Week 8,n=14,17 | 1.6 (7.76) | 3.4 (7.90)
  DBP, Week 12,n=10,12: number analyzed (Participants) | 10 | 12
  DBP, Week 12,n=10,12 | -1.0 (5.16) | 3.4 (7.01)
  DBP, Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  DBP, Week 16,n=7,7 | 0.7 (7.30) | 1.9 (9.56)
  DBP, Week 20,n=3,5: number analyzed (Participants) | 3 | 5
  DBP, Week 20,n=3,5 | 4.0 (0.00) | 5.6 (5.37)
  SBP, Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  SBP, Week 4,n=15,18 | 2.0 (8.99) | 2.6 (8.11)
  SBP, Week 8,n=14,17: number analyzed (Participants) | 14 | 17
  SBP, Week 8,n=14,17 | 0.6 (8.65) | 4.9 (11.24)
  SBP, Week 12,n=10,12: number analyzed (Participants) | 10 | 12
  SBP, Week 12,n=10,12 | -0.6 (6.62) | 2.8 (12.22)
  SBP, Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  SBP, Week 16,n=7,7 | 1.1 (5.76) | 3.3 (10.70)
  SBP, Week 20,n=3,5: number analyzed (Participants) | 3 | 5
  SBP, Week 20,n=3,5 | 0.7 (5.51) | 11.2 (6.14)

20. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Beats per minute
  Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  Week 4,n=15,18 | 0.3 (6.81) | 0.8 (9.80)
  Week 8,n=14,17: number analyzed (Participants) | 14 | 17
  Week 8,n=14,17 | 2.4 (9.57) | -1.4 (9.28)
  Week 12,n=10,12: number analyzed (Participants) | 10 | 12
  Week 12,n=10,12 | 0.6 (11.27) | 1.0 (12.41)
  Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  Week 16,n=7,7 | 3.7 (12.54) | -1.7 (15.68)
  Week 20,n=3,5: number analyzed (Participants) | 3 | 5
  Week 20,n=3,5 | 2.7 (5.86) | 0.8 (9.88)

21. Secondary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured in semi-supine position after 5 minutes rest for the participants at indicated time points. Day 1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and Weeks 4, 8, 12, 16 and 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Celsius
  Week 4,n=15,18: number analyzed (Participants) | 15 | 18
  Week 4,n=15,18 | 0.01 (0.474) | -0.02 (0.345)
  Week 8,n=14,17: number analyzed (Participants) | 14 | 17
  Week 8,n=14,17 | 0.06 (0.334) | 0.02 (0.281)
  Week 12,n=10,12: number analyzed (Participants) | 10 | 12
  Week 12,n=10,12 | 0.06 (0.357) | -0.29 (0.640)
  Week 16,n=7,7: number analyzed (Participants) | 7 | 7
  Week 16,n=7,7 | 0.14 (0.162) | -0.27 (0.309)
  Week 20,n=3,5: number analyzed (Participants) | 3 | 5
  Week 20,n=3,5 | -0.17 (0.153) | -0.08 (0.370)

22. Secondary Outcome: Number of Participants With Worst Post Baseline PCI Value for Vital Signs
Description: Blood samples were collected from participants for analysis of following vital signs parameters: DBP, Pulse rate and SBP. PCI ranges were <85 or >160 mmHg for SBP, <45 or >100 mmHg for DBP and < 40 or > 110 beats per minute for Pulse rate. Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there is no change in their category. Participants with vital signs value category "To Low" and "To High" were presented. Only those parameters having worst post-Baseline PCI values are presented. Day 1 was considered as Baseline.
Time Frame: Up to Week 20
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 18
Participants
  DBP,To Low | 0 | 0
  DBP,To High | 0 | 0
  Pulse rate, To Low | 0 | 0
  Pulse rate, To High | 0 | 1
  SBP,To Low | 0 | 0
  SBP,To High | 0 | 0

23. Secondary Outcome: Number of Participants With Abnormal Findings for ECG Parameters
Description: Triplicate 12-lead ECG were obtained to measure ECG parameters. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Week 4 and Week 16
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Participants
  Week 4; NCS; n=15, 18: number analyzed (Participants) | 15 | 18
  Week 4; NCS; n=15, 18 | 4 | 7
  Week 4; CS; n=15, 18: number analyzed (Participants) | 15 | 18
  Week 4; CS; n=15, 18 | 0 | 0
  Week 16; NCS; n= 12, 16: number analyzed (Participants) | 12 | 16
  Week 16; NCS; n= 12, 16 | 3 | 6
  Week 16; CS; n=12, 16: number analyzed (Participants) | 12 | 16
  Week 16; CS; n=12, 16 | 0 | 0

24. Secondary Outcome: Number of Participants With Any Time Post Baseline Anti-mepolizumab Binding Antibodies and Neutralizing Antibodies Response
Description: Blood samples were collected for the determination of anti-mepolizumab antibodies at the specified visits. The number of participants with anti-mepolizumab binding antibodies and neutralizing antibodies response at Any Time Post Baseline has been presented. Neutralizing antibodies response assay result have been only presented for participants with positive anti-drug antibody assay. Day 1 was considered as Baseline.
Time Frame: Up to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 19
Participants
  Binding Antibody, Negative, n=15,18: number analyzed (Participants) | 15 | 18
  Binding Antibody, Negative, n=15,18 | 15 | 17
  Binding Antibody, Positive, n=15,18: number analyzed (Participants) | 15 | 18
  Binding Antibody, Positive, n=15,18 | 0 | 1
  Neutralizing Antibody, Negative, n=0,1: number analyzed (Participants) | 0 | 1
  Neutralizing Antibody, Negative, n=0,1 | 0 | 1
  Neutralizing Antibody, Positive, n=0,1: number analyzed (Participants) | 0 | 1
  Neutralizing Antibody, Positive, n=0,1 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious Adverse events (SAEs) and nSAEs were collected from the start of study treatment Up to 20 weeks
Description: Safety Population was used. Safety Population comprised of all participants who received at least one dose of a study treatment. One participant from Placebo arm received Mepolizumab at Day 1 instead of placebo due to error.
Arm/Group | Placebo SC | Mepolizumab 100 mg SC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 7/15 | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SC (N=15) | Mepolizumab 100 mg SC (N=19)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03055195/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03055195/SAP_001.pdf